CLINICAL TRIAL: NCT06190808
Title: Continuous Glucose Monitoring in the Intensive Care Unit: Validation and Implementation
Brief Title: Continuous Glucose Monitoring in the Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, John P Mordes, MD, Professor Emeritus of Medicine, University of Massachusetts, Worcester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00001138
Record Dates: First submitted 2023-12-07; First posted 2024-01-05 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus
Keywords: ICU; CGM; Accuracy; Diabetes; Hypoglycemia; Diabetes mellitus; Continuous glucose monitor; Intensive care
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia

STUDY DESIGN:
Intervention Model Description: Hyperglycemic patients admitted to an intensive care unit will have blood glucose concentration measured using current standard-of-care tests (fingerstick determinations and laboratory assays). Study participants will bel be asked to volunteer to permit concurrent glucose measurement using a Dexcom G7 continuous glucose monitor in order to determine the accuracy and feasibility of the latter. Only standard glucose measurements will be used for patient management.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single Arm (Experimental): All members of the arm will have a CGM place and glucose concentration downloaded.
  Interventions: Diagnostic Test: Dexcom G7 Continuous Glucose Monitor

INTERVENTIONS:
Diagnostic Test: Dexcom G7 Continuous Glucose Monitor — Continuous glucose monitor

SUMMARY:
The aim of the proposed clinical trial is to study the use of the Dexcom G7 continuous glucose monitor (CGM) within the intensive care unit (ICU) environment. The overall goal is to validate the accuracy and practicality of the Dexcom G7 when used to assess glycemia in critically ill patients.

DETAILED DESCRIPTION:
The specific goals are 1) to work with intensive care unit (ICU) staff, in a respiratory ICU setting, to determine how best to place and maintain Dexcom G7 continuous glucose monitors (CGMs) on patients and how to place recording devices and chargers in that environment, 2) download CGM readings to the Dexcom Dashboard in an analyzable format, and 3) to compare simultaneous CGM readings with glucose measurements obtained in the course of routine care as recorded in the electronic medical record. The primary analytical goal is the correlation of CGM glucose measurements with those obtained in the course of routine care. A secondary goal is to determine the frequency of device malfunctions that occur either as a result of device failure (e.g. it falls off) or adverse events (e.g. removal due to skin irritation).

Study subjects will be patients admitted to the 6-ICU UMass Memorial Medical Center (UMMMC) University Campus medical intensive care unit for any reason who have known diabetes or who are hyperglycemic (blood glucose concentration ≥200 mg/dL) with diabetes that was previously undiagnosed or unrecognized. All enrolled volunteers will have a Dexcom G7 CGM place on the skin according to manufacturer's specifications. The devices will remain in place for 10 days or until discharge from the ICU

ELIGIBILITY:
Inclusion Criteria:

Campus medical intensive care unit for any reason who have known diabetes or who are hyperglycemic (blood glucose concentration ≥200 mg/dL) with diabetes that was previously undiagnosed or unrecognized.

* Persons with either type 1 or type 2 diabetes.
* Persons of either sex.
* Persons of any age over 18.
* Persons able to give informed consent or cognitively impaired adults whose legally authorized representative (LAR) can give informed consent.
* English or Spanish speaking adults.

Exclusion Criteria:

* Persons unable to provide informed consent.
* Cognitively impaired persons whose LAR declines to provide informed consent.
* Patients receiving hydroxyurea, which interferes with sensor function.
* Patients receiving high dose acetaminophen (> 4 gm/day), which interferes with sensor function.
* Anasarca affecting preferred areas for device placement (arm, upper buttocks, or thigh), which may interfere with sensor accuracy.
* Severe cachexia with absence of subcutaneous fat at preferred sensor placement sites, which might interfere with sensor accuracy.
* Persons who are pregnant.
* Prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Clarke Error Grid | 6 months
  Traditional comparison of glucose concentration results obtained by standard test methods and by newer method
Mean Absolute Relative Difference (MARD). | 6 months
  Concordance of glucose concentration results obtained by standard test methods with those obtained by a continuous glucose monitoring device

SECONDARY OUTCOMES:
Unplanned event frequency | 6 months
  Number of occurrences per patient of device failure or or unforeseen device removal
Adverse event nature and frequency | 6 months
  Number of occurrences per patient of device-associated infection, pain, or skin irritation

CONTACTS AND LOCATIONS:
Overall Officials: John P Mordes, MD, Principal Investigator — UMass Chan Medical School
Locations (1):
- UMass Memorial Medical Center, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Study design and deidentified aggregate glucose concentration data will be shared. No individual patient data will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: One year
Access Criteria: Publication